CLINICAL TRIAL: NCT01363232
Title: A Phase Ib, Open-label, Multi-center, Dose-escalation and Expansion Study of an Orally Administered Combination of BKM120 Plus MEK162 in Adult Patients With Selected Advanced Solid Tumors
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of BKM120 Plus MEK162 in Selected Advanced Solid Tumor Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162X2101; 2011-001083-22 (EudraCT Number)
Record Dates: First submitted 2011-05-24; First posted 2011-06-01 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Advanced Solid Tumors; Selected Solid Tumors
Keywords: BKM120; MEK162; RAS RAF mutations; triple negative breast cancer; pancreatic cancer, ovarian cancer; NSCLC progressed on EGFR TKI; PI3K inhibitor; MEK inhibitor
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms | interventions — NVP-BKM120; binimetinib

ARMS (1):
- BKM120 + MEK162 (Experimental)
  Interventions: Drug: BKM120 + MEK162

INTERVENTIONS:
Drug: BKM120 + MEK162

SUMMARY:
This is an open label, dose finding, phase Ib clinical trial to determine the maximum tolerated dose (MTD) and/or the recommended phase II dose (RP2D) of the orally administered phosphatidylinositol 3'-kinase (PI3K) inhibitor BKM120 in combination with the MEK1/2 inhibitor MEK162. This combination will be explored in patients with epidermal growth factor receptor (EGFR) mutant non-small cell lung cancer (NSCLC) which has progressed on EGFR inhibitors and triple negative breast cancer, as well as pancreatic cancer, colorectal cancer, malignant melanoma, NSCLC, and other advanced solid tumors with KRAS, NRAS, and/or BRAF mutations. Dose escalation will be guided by a Bayesian logistic regression model with overdose control. At MTD or RP2D, two expansion arms will be opened in order to further assess safety and preliminary anti-tumor activity of the combination of BKM120 and MEK162.

Study drugs will be administered once daily orally on a continuous schedule. A treatment cycle is defined as 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/ cytologically confirmed, advanced non resectable solid tumors
* Measurable or non-measurable, but evaluable disease as determined by RECIST

Exclusion Criteria:

* Patients with primary CNS tumor or CNS tumor involvement.
* Diabetes mellitus
* Unacceptable ocular/retinal conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | during Cycle 1 of treatment with BKM120 and MEK162

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events. | from Cycle 1 Day 1 until treatment discontinuation
Overall response rate, duration of response, time to response and progression free survival | every 8 weeks of treatment
Time versus plasma concentration profiles of BKM120 and MEK162 | during the first cycle of treatment on Cycle 1 Day 1 and Cycle 1 Day 15
Treatment -induced PI3K and MEK/ERK pathway signaling inhibition and evidence of biological activity in tumor. | during the first cycle of treatment on Cycle 1 Day 15 and at disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — 1-800-718-1021; Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (5):
  - Massachusetts General Hospital Mass General 2, Boston, Massachusetts
  - Karmanos Cancer Institute Study Coordinator, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center MSKCC (2), New York, New York
  - Cancer Centers of the Carolinas CCC Faris, Greenville, South Carolina
  - University of Texas/MD Anderson Cancer Center MD Anderson PSC, Houston, Texas
- Pfizer Investigative Site, Toronto, Ontario, Canada
- Germany (2):
  - Pfizer Investigative Site, Essen
  - Pfizer Investigative Site, Heidelberg
- Pfizer Investigative Site, Utrecht, Netherlands
- Pfizer Investigative Site, Singapore, Singapore
- Pfizer Investigative Site, Barcelona, Catalonia, Spain
- Pfizer Investigative Site, Bellinzona, Switzerland

REFERENCES:
- [Derived] Bardia A, Gounder M, Rodon J, Janku F, Lolkema MP, Stephenson JJ, Bedard PL, Schuler M, Sessa C, LoRusso P, Thomas M, Maacke H, Evans H, Sun Y, Tan DSW. Phase Ib Study of Combination Therapy with MEK Inhibitor Binimetinib and Phosphatidylinositol 3-Kinase Inhibitor Buparlisib in Patients with Advanced Solid Tumors with RAS/RAF Alterations. Oncologist. 2020 Jan;25(1):e160-e169. doi: 10.1634/theoncologist.2019-0297. Epub 2019 Aug 8. PMID 31395751